CLINICAL TRIAL: NCT05158179
Title: Assessment of Laryngopharyngeal Sensation in Adductor Spasmodic Dysphonia
Acronym: SDTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Spasmodic Dysphonia Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB: 20-31653
Record Dates: First submitted 2021-11-18; First posted 2021-12-15 (Actual); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Spasmodic Dysphonia; Adductor Spasmodic Dysphonia; Voice Disorders
Keywords: throat sensation
MeSH Terms: conditions — Dysphonia; Voice Disorders

STUDY DESIGN:
Intervention Model Description: Cottonoid pledgets soaked in 4% lidocaine and neo-synephrine will be placed on this side. The pledgets will be kept in place for 5 minutes to allow adequate decongestion and anesthetization. The aesthesiometer will be placed through the 2.0 mm working channel of the Olympus Corporation (Tokyo, Japan) ENF-VT2 channeled flexible video rhinolaryngoscope with a 4.9 mm outer diameter. The flexible laryngoscope and aesthesiometer assembly will then be advanced into the pharynx and positioned for target testing. The operator field of view will be adjusted in the craniocaudal axis to optimize visualization of the stimulation target, monofilament tip, and both vocal folds to assess for a stimulation evoked LAR response. The monofilament will then be advanced to within several mm of the target laryngopharyngeal subsite and subsequently applied orthogonally until it buckled by 10-30%, followed by quick retraction to assess for triggering of the rapid LAR response.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Spasmodic Dysphonia Patients (Experimental): Following appropriate nasal local anesthetic, the channeled laryngoscope was inserted through the nose. The 6-0 monofilament was pressed against the posterior nasopharyngeal wall and swiftly removed to establish a perceptual strength of "1", as an internal anchor. The lateral pyriform sinus (LPS) was presented with the planned stimulus, followed by the aryepiglottic fold (AEF) and the false vocal folds (FVF). Participants were instructed to raise their hand when the stimulus was detected, and then were asked by the study team to report a perceptual strength "score," in comparison to the nasopharyngeal anchor strength of 1. LAR response was recorded by the study team. A negative response was defined as a lack of LAR to two appropriate stimuli. The LPS and AEF were tested in order of increasing stimulus: 6-0, 5-0, 4.5-0 and 4-0 monofilaments. The false vocal folds (FVF) were tested last. Testing of FVF terminated after the first observed LAR.
  Interventions: Device: Sensation testing

INTERVENTIONS:
Device: Sensation testing — Sensation testing tactile aesthesiometer.

SUMMARY:
Study investigators have completed a study testing laryngopharyngeal sensation at specific laryngopharyngeal subsites using a novel buckling force aesthesiometer in a series of 22 healthy adults at this institution. Investigators would like to use the same device apparatus to evaluate laryngopharyngeal sensation in patients with laryngopharyngeal disorders, such as adductor spasmodic dysphonia. This study will use a tested laryngopharyngeal aesthesiometer to examine laryngeal sensation using calibrated tactile stimuli to determine differences in somatotopic perceptual strength maps of laryngopharyngeal structures between patients with laryngopharyngeal disorders and healthy controls.

DETAILED DESCRIPTION:
Participant Recruitment Subjects with adductor type LD (AdLD) were identified and recruited by advertisements and by study clinicians at their institution. Advertisements were physically placed in the UCSF Voice and Swallowing Center clinic and were delivered electronically through the website of the National Spasmodic Dysphonia Association and to area LD ("spasmodic dysphonia") support groups.

Adults greater than 18 years old with AdLD were included if they received a diagnosis established by a multi-disciplinary evaluation by a fellowship-trained laryngologist and voice-specialized speech-language pathologist. Subjects diagnosed by a physician outside of the study facility were evaluated in-person by a fellowship-trained laryngologist to confirm their eligibility for this study. All patients were required to have history of favorable response to intra-laryngeal botulinum toxin A (BtxA) treatment, as further demonstration of the correct diagnosis of ADLD. This was especially helpful for patients initially diagnosed outside of our center. Subjects with abductor or mixed type LD were not included in the present study due to their low incidence, but concurrent essential tremor (ET) of the vocal tract was accepted.

Patients were also excluded if they had a history of: concurrent laryngeal diseases or conditions other than AdLD+/-ET; bleeding disorder or current anticoagulation use; head and neck radiation; active tobacco use; or drinking more than two alcoholic beverages per day. If laryngopharyngeal lesions and/or masses, impeding abnormal laryngopharyngeal structure(s), or excessive post-nasal drip were noted on laryngoscopy, then examination ceased, and patients were excluded. Prior to testing, subjects also completed symptom-specific patient reported outcome measures (PROMs), including: Reflux Symptom Index (RSI),18 Voice Handicap Index-10 (VHI-10),19 Dyspnea Index (DI),20 Cough Severity Index (CSI),21 and Eating Assessment Tool-10 (EAT-10).22 These PROMs are standardly collected as part of the routine clinical are for all patients undergoing evaluation at this center and are reported herein for holistic characterization of these subjects but not intended as a reflection or measure of the severity of their AdLD. Lastly, to avoid any potentially confounding physical effects from the injection (e.g., vocal fold edema), no testing was performed in the two weeks immediately following BtxA treatment. For patient convenience and to facilitate maximal enrollment, patients were allowed to undergo testing at any point outside of this post-injection window, although the majority pursued testing immediately prior to a BtxA injection on the same day.

Healthy controls were defined as adults between 18 and 85 years of age without laryngopharyngeal disease and were subject to the same screening and exclusion criteria.23 Additionally, controls were excluded if they had abnormal patient reported outcome measures (i.e. Reflux Symptom Index (RSI) score> 13, Eating Assessment Tool-10 (EAT-10) score>2, or Voice Handicap Index-10 (VHI-10) score> 11).

Aesthesiometer Device As outlined in previous work, modified nylon monofilaments fixed to the end of 5-French open lumen catheters were utilized to deliver tactile stimuli to laryngopharyngeal subsites.12 The Food and Drug Administration (FDA) has previously ruled the aesthesiometer to be a Nonsignificant Risk (NSR) Device Study (Q190371/S001). Three nylon monofilament sizes (6-0, 5-0, 4-0) were cut to a calibrated length of 30 mm to deliver three distinct tactile stimuli of increasing strength, known as buckling-force. The 6-0, 5-0, and 4-0 monofilaments deliver an increasing mean force of 0.03 g, 0.11 g, and 0.30 g, respectively.12 An intermediary strength "4.5-0" monofilament was created by using a 5-0 monofilament of 25mm length, which has been demonstrated to have a mean buckling force of 0.19 g.23 During testing, the monofilaments were passed through the working channel of a flexible ENF-VT2 laryngoscope (Olympus America, Inc., Center Valley, PA) to allow for direct visualization and concurrent stimulation of laryngopharyngeal subsites.

Laryngopharyngeal Sensory Evaluation All subjects underwent a standard protocol for laryngopharyngeal sensory evaluation. This has been described in detail previously but briefly reviewed again here.12,13 Prior to testing, subjects were screened for any recent changes in conditions affecting voice and swallowing to ascertain subjects-maintained inclusion criteria. Three investigators executed laryngopharyngeal testing: 1) one to operate the laryngoscope; 2) one to maneuver the aesthesiometer monofilament; and 3) one to monitor testing, record subjective patient response, and observe cough/gag/swallow responses.

An investigator then examined both nasal passageways with a nasal speculum, selecting the more patent pathway for laryngoscope insertion. The more patent nasal passageway was topically anesthetized with cottonoid pledgets soaked in a 50/50 mixture of 4% lidocaine hydrochloride and neosynephrine. The cottonoid pledgets were compressed to remove excess liquid to avoid unintentional spillage posteriorly to the nasopharynx and potentially larynx, and left in place for five minutes.

The channeled laryngoscope was then inserted along the inferior meatus towards the posterior nasopharyngeal wall. The 6-0 monofilament was pressed against the posterior nasopharyngeal wall and swiftly removed to establish a perceptual strength of "1". If subjects were insensate to this stimulation, monofilament size was incrementally increased (i.e., 5-0, 4.5-0, and 4-0) until the stimulus was perceived, to establish this internal anchor. As per the validated, standardized protocol, all AdLD participants were stimulated on the left, allowing maximal visualization of the vocal folds during testing due to camera configuration of the flexible laryngoscope. Only four controls were stimulated on the right side, during earliest phases of testing.

Starting with the 6-0 monofilament, the lateral pyriform sinus (LPS) was presented with the planned stimulus, followed by the aryepiglottic fold (AEF) and the false vocal folds (FVF). (Figure 1) Participants were instructed to raise their hand when the stimulus was detected, and then were asked by the study team to report a perceptual strength "score," in comparison to the nasopharyngeal anchor strength of 1. LAR response was observed and recorded by the study team. A negative response was defined as a lack of LAR to two appropriate stimuli. Gag or cough response to stimuli delivery were also recorded, assuming a positive LAR during these observations.

The LPS and AEF were tested in order of increasing stimulus: 5-0, 4.5-0 and 4-0 monofilaments. The false vocal folds (FVF) were tested last, in the same order of increasing monofilament strength. Testing of FVF terminated after the first observed LAR given site sensitivity, assuming positive responses would also be present for increased monofilament strength.

LAR Assessment Confirmation of LAR was determined using post-hoc frame-by-frame analysis of video recordings. Unilateral or bilateral vocal fold adduction following stimulus delivery was recorded as a positive response. Upon review, stimuli were excluded if they did not produce 10-30% monofilament buckling (as observed by the reviewer), were entrapped by saliva, or could not compress orthogonally to the mucosal surface. Additionally, if line of sight of visualization of vocal fold adduction was obstructed or confounded by phonation, the stimuli were excluded. All stimuli were reviewed by one study investigator with 30% of stimuli reviewed by a blinded second reviewer. Disagreements were reconciled by a blinded third reviewer.

ELIGIBILITY:
Inclusion Criteria:

* Adductor spasmodic dysphonia (can have co-diagnosis of essential tremor)
* received Botox injection more than 2 weeks ago

Exclusion Criteria:

* excessive gagging
* active smoker
* non-Botox responsive
* abductor spasmodic dysphonia exclusively
* essential tremor diagnosis exclusively

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yue Ma, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Voice and Swallowing Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bearelly S, Cheung SW. Sensory Topography of Oral Structures. JAMA Otolaryngol Head Neck Surg. 2017 Jan 1;143(1):73-80. doi: 10.1001/jamaoto.2016.2772. PMID 27684535
- [Background] Bearelly S, Wang SJ, Cheung SW. Oral sensory dysfunction following radiotherapy. Laryngoscope. 2017 Oct;127(10):2282-2286. doi: 10.1002/lary.26591. Epub 2017 Apr 11. PMID 28397276
- [Background] Aviv JE, Martin JH, Keen MS, Debell M, Blitzer A. Air pulse quantification of supraglottic and pharyngeal sensation: a new technique. Ann Otol Rhinol Laryngol. 1993 Oct;102(10):777-80. doi: 10.1177/000348949310201007. PMID 8215097
- [Background] Aviv JE, Martin JH, Kim T, Sacco RL, Thomson JE, Diamond B, Close LG. Laryngopharyngeal sensory discrimination testing and the laryngeal adductor reflex. Ann Otol Rhinol Laryngol. 1999 Aug;108(8):725-30. doi: 10.1177/000348949910800802. PMID 10453777
- [Background] Strohl MP, Young VN, Dwyer CD, Bhutada A, Crawford E, Chang JL, Rosen CA, Cheung SW. Novel Adaptation of a Validated Tactile Aesthesiometer to Evaluate Laryngopharyngeal Sensation. Laryngoscope. 2021 Jun;131(6):1324-1331. doi: 10.1002/lary.28947. Epub 2020 Jul 31. PMID 32735711

RESULTS

PARTICIPANT FLOW:
Groups:
- Spasmodic Dysphonia Patients: Patients with Spasmodic Dysphonia underwent one-time testing of laryngeal sensation using a validated methodology involving a tactile esthesiometer. Various sizes of monofilament device were passed through the working channel of a flexible laryngoscope passed through the nose under local anesthesia. This study involved SD patients to then be compared to historical controls already assessed previously at our institution.
Period: Overall Study
Arm/Group | Spasmodic Dysphonia Patients
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Spasmodic Dysphonia Patients: Sensation testing of Spasmodic Dysphonia Patients
Arm/Group | Spasmodic Dysphonia Patients
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13
Voice Handicap Index-10 (VHI-10) [Mean (Standard Deviation); unit: units on a scale] — The Voice Handicap Index-10 (VHI-10) is a questionnaire involving 10 items, scored from 0-4. Scores are reported as cumulative total. Total score ranges from 0-40, with higher scores indicating greater patient-reported voice-related handicap.
  units on a scale | 24 (9.4)

OUTCOME MEASURES:

1. Primary Outcome: Laryngeal Adductor Reflex
Description: The outcome measure is the presence or absence of a laryngeal adductor reflex (LAR) which is the reflexive, involuntary closure of the vocal folds in response to stimulation, as seen on flexible laryngoscopy. This is a binary finding in that this is immediately observed as either being present or absent following direct contact by the tactile esthesiometer device. Accordingly, there are no units of measure. The presence or absence of the LAR was noted at the time of testing by the study team and confirmed on subsequent video review by another member of the study team. This study only examined patients with SD - all of whom were found to have LAR present.
Time Frame: Immediately after intervention, less than 10 seconds
Measure: Count of Participants; unit: Participants
Arm/Group | Spasmodic Dysphonia Patients
Number analyzed (Participants) | 13
Participants | 13

2. Secondary Outcome: Perceptual Strength of Sensation on a 1-10 Numerical Rating Scale (NRS)
Description: The smallest size tactile aesthesiometer was utilized to establish an internal anchor base score of 1 based on direct palpation of the posterior nasopharyngeal wall. Participants were instructed to rate all subsequent perceptual strength testings in comparison to this individualized, internal anchor. During testing, participants were instructed to raise their hand when the stimulus was detected, and then were asked by the study team to report a perceptual strength "score" from 1-10, in comparison to the nasopharyngeal anchor strength of 1, with 1 being the same as the barest perception of touch within the nasopharynx and 10 being 10-fold stronger sensation. It was not anticipated that any perceived sensation within the larynx (a more sensitive organ than the nasopharynx) would be lower than the lowest perceived sensation in the nose.
Time Frame: Immediately after intervention, within 30 seconds
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spasmodic Dysphonia Patients
Number analyzed (Participants) | 13
units on a scale | 4.6 (2.8)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at the time of the testing including 10 minutes after conclusion of testing.
Description: Patients were directly observed by the study team including a board certified otolaryngologist during and immediately after the procedure. Any adverse events - either major or minor - were documented by the study team.
Arm/Group | Spasmodic Dysphonia Patients
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT05158179/Prot_SAP_001.pdf